CLINICAL TRIAL: NCT01177293
Title: Phase 1, Open-Label, Randomized, Single-Dose, 2-Treatment, 2-Period Crossover Bioavailability Study Comparing 10 Mg Amlodipine Besylate Orally Disintegrating Tablets, Manufactured By Aurobindo Pharma Ltd., India To 10 Mg Amlodipine Besylate Capsules, Manufactured By Pfizer France Under Fasted Conditions
Brief Title: Bioavailability Study Comparing 10 mg Amlodipine Besylate Orally Disintegrating Tablets (ODT) And 10 mg Amlodipine Besylate Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Aurobindo Pharma Ltd (Industry); Trident Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0531096; 052-10
Record Dates: First submitted 2010-03-10; First posted 2010-08-06 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: biological availability; bioavailability; amlodipine; orally disintegrating tablet; ODT; tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment A - reference w/ water (Active Comparator)
  Interventions: Drug: Amlodipine - reference
- Treatment B - ODT (test) w/o water (Experimental)
  Interventions: Drug: Amlodipine ODT - test

INTERVENTIONS:
Drug: Amlodipine - reference — Amlodipine capsule, 10 mg, single dose, with water
  Arms: treatment A - reference w/ water
Drug: Amlodipine ODT - test — Amlodipine orally disintegrating tablet (ODT), 10 mg, single dose, without water
  Arms: Treatment B - ODT (test) w/o water

SUMMARY:
This study is being performed to determine the bioavailability, or extent of absorption into the body, of a 10 mg amlodipine besylate orally disintegrating tablet (ODT) as compared to the bioavailability of a 10 mg amlodipine besylate capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female literate subjects (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 26.4 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hydrabad, Andhra Pradesh, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531096&StudyName=Bioavailability%20Study%20Comparing%2010%20mg%20Amlodipine%20Besylate%20Orally%20Disintegrating%20Tablets%20%28ODT%29%20And%2010%20mg%20Amlodipine%20Besylate%20Capsules

RESULTS

PARTICIPANT FLOW:
Groups:
- Amlodipine Capsule Then Amlodipine ODT: Single oral dose amlodipine besylate 10 mg capsule in first intervention period and single oral dose of amlodipine besylate 10 mg oral disintegrating tablet (ODT) in second intervention period. A washout period of 14 days was maintained between each period.
- Amlodipine ODT Then Amlodipine Capsule: Single oral dose amlodipine besylate 10 mg ODT in first intervention period and single oral dose of amlodipine besylate 10 mg capsule in second intervention period. A washout period of 14 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Amlodipine Capsule Then Amlodipine ODT | Amlodipine ODT Then Amlodipine Capsule
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period (of 14 Days)
Arm/Group | Amlodipine Capsule Then Amlodipine ODT | Amlodipine ODT Then Amlodipine Capsule
Started | 7 | 7
Completed | 7 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention Period
Arm/Group | Amlodipine Capsule Then Amlodipine ODT | Amlodipine ODT Then Amlodipine Capsule
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive any treatment first (amlodipine capsule first and amlodipine ODT first).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.00 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 and 168 hours post dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Full Range); unit: hr*ng/mL
Groups:
- Amlodipine 10 mg Capsule: Single oral dose of amlodipine 10 mg capsule (Treatment A [Reference]).
- Amlodipine 10 mg ODT: Single oral dose of amlodipine 10 mg ODT (Treatment B [Test]).
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Number analyzed (Participants) | 12 | 13
hr*ng/mL | 401.655 [61.74 to 566.54] | 360.619 [266.76 to 635.54]
Statistical Analysis 1: Comparison: Amlodipine 10 mg Capsule vs Amlodipine 10 mg ODT; A sample size of 12 completers provided 90% confidence intervals for the difference between treatment of +/-0.1155 on the natural log scale for AUCinf with 90% coverage probability. These calculations were based on estimates of within-participant standard deviations of 0.1234 for loge AUCinf; Test type: Non-Inferiority or Equivalence — Natural log transformed AUC[0- ∞] of amlodipine was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect.The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Adjusted geometric means ratio = 89.78, 90% CI 2-sided [82.74 to 97.43]

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration-time curve from time zero (pre-dose) to the time of the last measurable concentration (AUClast).
Time Frame: 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 and 168 hours post dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Full Range); unit: hr*ng/mL
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Number analyzed (Participants) | 12 | 13
hr*ng/mL | 331.300 [60.42 to 463.69] | 330.394 [243.87 to 558.60]
Statistical Analysis 1: Comparison: Amlodipine 10 mg Capsule vs Amlodipine 10 mg ODT; Test type: Non-Inferiority or Equivalence — Natural log transformed AUClast of amlodipine was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect.The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Adjusted geometric mean ratio = 99.73, 90% CI 2-sided [85.10 to 116.87]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 and 168 hours post dose
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Number analyzed (Participants) | 12 | 13
ng/mL | 6.427 [1.88 to 8.32] | 5.571 [3.92 to 7.84]
Statistical Analysis 1: Comparison: Amlodipine 10 mg Capsule vs Amlodipine 10 mg ODT; A sample size of 12 completers provided 90% confidence intervals for the difference between treatment of +/-0.1278 on the natural log scale for Cmax with 90% coverage probability. These calculations were based on estimates of within-participant standard deviations of 0.1366 for loge Cmax; Test type: Non-Inferiority or Equivalence — Natural log transformed Cmax of amlodipine was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Adjusted geometric means ratio = 86.67, 90% CI 2-sided [79.57 to 94.42]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 and 168 hours post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Number analyzed (Participants) | 12 | 13
hr | 8.00 [6.00 to 14.00] | 10.00 [6.00 to 14.00]

5. Secondary Outcome: Plasma Decay Half-life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 and 168 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Number analyzed (Participants) | 12 | 13
hr | 51.374 (12.912) | 45.120 (4.921)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Amlodipine 10 mg Capsule | Amlodipine 10 mg ODT
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.